CLINICAL TRIAL: NCT05874180
Title: A Phase 1 Clinical Trial to Compare and Evaluate the Safety and Pharmacokinetic Characteristics After Administration of Fixed-dose Combination of DW6013 and Loose Combination of Each Component in Healthy Adult Volunteers in Fed Condition
Brief Title: A Pharmacokinetic Study of DW6013 (FDC of Linagliptin and Metformin) in Healthy Adult Volunteers in Fed Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong Wha Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW6013-I-2
Record Dates: First submitted 2023-04-06; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Jentadueto

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental): Period 1: Linagliptin and Metformin / Period 2: DW6013
  Interventions: Drug: DW6013
- Sequence B (Experimental): Period 1: DW6013 / Period 2: Linagliptin and Metformin
  Interventions: Drug: DW6013

INTERVENTIONS:
Drug: DW6013 — Drug: DW6013 Single oral administration of DW6013 in fed condition
  Drug: Linagliptin and Metformin Single oral administration of Linagliptin and Metformin in fed condition
  Other Names: Linagliptin and Metformin

SUMMARY:
This study is to compare and evaluate the safety and pharmacokinetic characteristics (PK) after administration of DW6013 and each component in healthy adult volunteers in fed condition.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, open-label, Oral, Single-dose, two-way crossover study in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged up to 19 years
* Subjects weighing at least 50.0 kg and no more than 100 kg (inclusive) with a BMI between 18.5 kg/m2 and 30.0 kg/m2
* Subjects with neither congenital nor chronic diseases requiring treatment, and no abnormal symptoms or findings upon medical examination
* Subjects considered eligible for the study participation in accordance to the results of clinical laboratory tests, vital signs, physical examinations and 12-lead ECG conducted at the time of screening, based on the investigational product (IP) characteristics
* Subjects who has a full understanding in participation of the study, voluntarily provide a written consent in participation, and give full agreement in following the subject guidelines throughout the entire study period

Exclusion Criteria:

* Subjects with any clinically significant hepatic, renal, nervous, respiratory, endocrine, circulatory, tumor, genitourinary, cardiovascular, digestive, musculoskeletal systemic diseases or other medical history
* Pregnant subjects with a positive urine HCG test, or lactating female subjects
* Subjects taking drugs known to significantly induce or inhibit drug metabolizing enzymes, including barbitals within 1 months prior to the first IP administration
* Subjects with clinically significant 12-lead ECG findings at the time of screening
* Subjects with a past history of drug abuse or a positive urine drug test
* Subjects with SBP ≥ 150 mmHg or ≤ 90 mmHg; DBP ≥ 100 mmHg or ≤ 60 mmHg; PR ≤ 40 bpm or ≥ 100 bpm at the time of screening
* Subjects following an unusual diet or consumption of food which may affect the absorption, distribution, metabolism and excretion of the IP
* Subjects who have administered any prescription drugs or herbal medicines that may affect the characteristics of clinical investigational drugs within 2 weeks prior to the first administration date, or have administered any over-the-counter (OTC) or vitamin preparations within 10 days
* Subjects who have participated and were given any other study drugs in other clinical study within 6 months prior to the first IP administration
* Subjects who have consistently drunk alcohol within 6 months
* Subjects who have smoked more than 10 cigarettes/day on average
* Subjects who have eaten or cannot refrain from eating grapefruit (grapefruit)-containing food from 48 hours before the first administration until the time of PSV
* Subjects who have consumed or cannot refrain from consuming caffeine-containing food during the period from 24 hours prior to administration of each period to the time of the last blood sampling
* Subjects who have done and are unable to refrain from strenuous activity
* Subjects who are planning for pregnancy or not willing to use a medically reliable forms of contraception
* Subjects otherwise considered ineligible for participation due to other reasons including clinical laboratory test results not mentioned in the inclusion/exclusion criteria at the investigator's discretion

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
AUC0-t | up to 48 hours
  AUC0-t of Metformin
Cmax | up to 48 hours
  Cmax of Metformin

SECONDARY OUTCOMES:
Tmax | up to 48 hours
  Tmax of Metformin
AUCinf | up to 48 hours
  AUCinf of Metformin
t1/2 | up to 48 hours
  t1/2 of Metformin
CL/F | up to 48 hours
  CL/F of Metformin
Vd/F | up to 48 hours
  Vd/F of Metformin

CONTACTS AND LOCATIONS:
Locations (1):
- Chungbuk National University Hospital, Cheongju-si, South Korea

IPD SHARING:
Plan to Share IPD: No